CLINICAL TRIAL: NCT02539719
Title: A Phase 1a/1b Dose Escalation and Expansion Study of SC-003 as a Single-Agent and in Combination With ABBV-181 in Subjects With Platinum-Resistant/ Refractory Ovarian Cancer
Brief Title: Study of SC-003 Alone and in Combination With ABBV-181 in Subjects With Platinum-Resistant/Refractory Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Considerations
Sponsor: Stemcentrx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCRX003-001
Record Dates: First submitted 2015-08-26; First posted 2015-09-03 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer
Keywords: Platinum-Resistant; Refractory
MeSH Terms: conditions — Ovarian Neoplasms | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SC-003 (Experimental): Phase 1a (Escalation) - IV infusion Phase 1b (Expansion) - IV infusion
  Interventions: Drug: SC-003
- SC-003 in combination with ABBV-181 (Experimental): Phase 1a (Escalation) - IV infusion of SC-003 followed by IV infusion of ABBV-181 Phase 1b (Expansion) - IV Infusion of SC-003 followed by IV infusion of ABBV-181
  Interventions: Drug: SC-003 in combination with ABBV-181

INTERVENTIONS:
Drug: SC-003
  Arms: SC-003
Drug: SC-003 in combination with ABBV-181
  Arms: SC-003 in combination with ABBV-181

SUMMARY:
This is a Phase 1a/1b study of SC-003 as a single agent and in combination with ABBV-181 in patients with platinum-resistant/refractory ovarian cancer. SC-003 is an antibody-drug conjugate (ADC) comprised of a monoclonal antibody linked to a potent chemotherapy. ABBV-181 is a humanized, recombinant, mAb that binds to cell surface expressed programmed cell death 1 (PD-1).

DETAILED DESCRIPTION:
Phase 1a is a dose escalation study in patients with histologically/cytologically confirmed ovarian cancer that are platinum-resistant or refractory. Phase 1b is an expansion study where patients will be enrolled and treated at recommended dose and schedule based on the Phase 1a.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ovarian epithelial cancer
* Evidence of progressive disease (PD) on or within 6 months of a platinum (cisplatin or carboplatin) regimen: at least 1 prior regimen must have contained a platinum-taxane combination
* Measurable disease as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Fresh or archived tumor tissue sample available for target expression analysis. [Phase 1b only: Subjects' tumor tissue must test positive for target expression.]
* Adequate hematologic and organ function as confirmed by laboratory values
* At least 3 weeks between last systemic chemotherapy and planned start of study treatment (4 weeks for prior investigational drugs, immunotherapy, radiotherapy, or biologics) for ovarian cancer
* At least 3 weeks between major surgery and planned start of study treatment; major incisions must have healed

Exclusion Criteria:

* History of prior malignancy, with the exception of the following: malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening and felt to be at low risk for recurrence by treating physician; or adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer; or adequately treated cervical carcinoma in situ without current evidence of disease.
* Uncontrolled infection requiring systemic antibiotics/antivirals/antifungals
* Evidence of complete or partial bowel obstruction
* Patients requiring IV hydration or parenteral nutrition
* Positive pregnancy test in females of child-bearing potential or pregnant or currently breastfeeding
* Known hypersensitivity to any component of study drug including potential subjects with a history of major immunologic reaction to any IgG-containing agent
* Inability to tolerate premedication with dexamethasone
* Uncontrolled cardiac disease, or myocardial infarction within the last 12 months, or left ventricular ejection fraction (LVEF) < 50%, or QTcF interval > 470 msec
* Class II, III or IV heart failure as defined by the NYHA functional class system
* Positive serology for hepatitis B or C, or known human immunodeficiency virus infection (HIV)
* Previous treatment with a pyrrolobenzodiazepine (PBD)-based drug

Additional exclusion criteria for the SC-003 and ABBV-181 combination treatment regimen:

* History of inflammatory bowel disease
* Active autoimmune disease, with exceptions of psoriasis not requiring systemic treatment, vitiligo, type 1 diabetes mellitus and hypothyroidism
* History of primary immunodeficiency, allogeneic bone marrow transplantation, solid organ transplantation, or previous clinical diagnosis of tuberculosis
* History of immune-mediated pneumonitis
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 18 months (Phase 1a/1b)

SECONDARY OUTCOMES:
Overall Response Rate | 18 months (Phase 1a/1b)
Pharmacokinetics of SC-003: AUC (area under the curve) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min)
Pharmacokinetics of SC-003: Cmax (maximum concentration) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min
Pharmacokinetics of SC-003: Tmax (time of maximum concentration) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min
Pharmacokinetics of SC-003: Ctrough (concentration at trough) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min
Pharmacokinetics of SC-003: T1/2 (terminal half life) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min
Pharmacokinetics of SC-003: CL (clearance) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min
Pharmacokinetics of SC-003: Vss (volume of distribution at steady state) | Cycle 1 and 4: days 1 (pre-dose, post-dose: 30min, 6hr), 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 (pre-dose, post-dose: 30min

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lawrence, D.O., Study Director — Novella Clinical
Locations (15):
- United States (15):
  - Fayetteville, Arkansas
  - Duarte, California
  - Chicago, Illinois
  - Evanston, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Hamilton E, O'Malley DM, O'Cearbhaill R, Cristea M, Fleming GF, Tariq B, Fong A, French D, Rossi M, Brickman D, Moore K. Tamrintamab pamozirine (SC-003) in patients with platinum-resistant/refractory ovarian cancer: Findings of a phase 1 study. Gynecol Oncol. 2020 Sep;158(3):640-645. doi: 10.1016/j.ygyno.2020.05.038. Epub 2020 Jun 6. PMID 32513564